CLINICAL TRIAL: NCT00824499
Title: Development, Implementation and Evaluation of a Complex Regional Intervention for Type 2 Diabetes.
Brief Title: Development, Implementation and Evaluation of a Complex Regional Intervention for Type 2 Diabetes: Diabetes Project Aalst
Acronym: DPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Belgian National Health Insurance Organisation (RIZIV) (Unknown); University Ghent (Other)
Responsible Party: Prof.dr. Paul Van Royen, Department of General Practice, University of Antwerp
Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A0456
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DPA (Experimental): Regional complex intervention based on the Chronic Care Model
  Interventions: Other: Complex regional intervention
- VR (No Intervention)

INTERVENTIONS:
Other: Complex regional intervention — Components of the complex intervention:
  * Introduction of a program coordinator
  * Introduction of a self-management education program
  * Bottom up development of a interdisciplinary care protocol
  * Support program for the intiation of insulin therapy in primary care
  * Regional audit
  Arms: DPA

SUMMARY:
The purpose of this study is to determine whether regional implementation of shared care with respect to type 2 diabetes is feasible, effective and cost-effective.

DETAILED DESCRIPTION:
Background Diabetes is an important chronic condition with significant associated morbidity and mortality, which can be reduced by effective care. An interdisciplinary approach, sharing responsibility and involvement and education of patients are of major importance in diabetes care.

In Belgium a research project aimed at creating regional diabetes shared care was set up.

Research questions

* Is regional implementation of shared care feasible?
* Does it increases quality of care (evidence based care) and patient satisfaction with care?
* Does it have a positive effect on health status (emotional distress, overall quality of life, Hba1c)?

Methods Controlled trial (July 2004 - June 2006) with a regional complex intervention comprising introduction of a care-manager and 2 community based diabetes educators, development and implementation of a shared care protocol (with a central role for the GP), regional feedback on the quality of diabetes care and patient education. Practitioners and patients participate on a voluntary basis. In the control region usual care continues.

Biophysical, psychosocial and process outcomes were collected thru GP registration of patients records and self-administered patient questionnaires (PAID, QUOTE).

ELIGIBILITY:
Inclusion Criteria:

* All type 2 diabetes patients living in the defined intervention region
* All caregivers involved in type 2 diabetes care in the defined intervention region

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2004-02; Primary Completion 2007-12 (Actual); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
HBA1C | Longitudinal analysis on measurements from 01/01/2004 until 31/12/2006

SECONDARY OUTCOMES:
Total Cholesterol | Longitudinal analysis on measurements from 01/01/2004 until 31/12/2006
LDL-C | Longitudinal analysis on measurements from 01/01/2004 until 31/12/2006
HDL-C | Longitudinal analysis on measurements from 01/01/2004 until 31/12/2006
microalb. | Longitudinal analysis on measurements from 01/01/2004 until 31/12/2006
blood creatinine | Longitudinal analysis on measurements from 01/01/2004 until 31/12/2006
ophthalmist consults | Longitudinal analysis on measurements from 01/01/2004 until 31/12/2006
Statine prescriptions | Longitudinal analysis on measurements from 01/01/2004 until 31/12/2006
Influenza Vaccination Prescriptions | Longitudinal analysis on measurements from 01/01/2004 until 31/12/2006

CONTACTS AND LOCATIONS:
Overall Officials: Paul Van Royen, Prof. Ph.D. M.D., Study Director — Universiteit Antwerpen; Jan De Maeseneer, Prof. Ph.D. M.D., Study Director — University Ghent

REFERENCES:
- [Derived] Sunaert P, Willems S, Feyen L, Bastiaens H, De Maeseneer J, Jenkins L, Nobels F, Samyn E, Vandekerckhove M, Wens J, De Sutter A. Engaging GPs in insulin therapy initiation: a qualitative study evaluating a support program in the Belgian context. BMC Fam Pract. 2014 Aug 21;15:144. doi: 10.1186/1471-2296-15-144. PMID 25145469
- [Derived] Sunaert P, Bastiaens H, Nobels F, Feyen L, Verbeke G, Vermeire E, De Maeseneer J, Willems S, De Sutter A. Effectiveness of the introduction of a Chronic Care Model-based program for type 2 diabetes in Belgium. BMC Health Serv Res. 2010 Jul 14;10:207. doi: 10.1186/1472-6963-10-207. PMID 20630062
- [Derived] Sunaert P, Bastiaens H, Feyen L, Snauwaert B, Nobels F, Wens J, Vermeire E, Van Royen P, De Maeseneer J, De Sutter A, Willems S. Implementation of a program for type 2 diabetes based on the Chronic Care Model in a hospital-centered health care system: "the Belgian experience". BMC Health Serv Res. 2009 Aug 23;9:152. doi: 10.1186/1472-6963-9-152. PMID 19698185